CLINICAL TRIAL: NCT01264978
Title: Evaluation of Utility Quadriceps Magnetic Stimulation in COPD (Chronic Obstructive Pulmonary Disease) Patients After Hospital Exacerbation
Acronym: COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Cruces (Other)
Collaborators: Basurto hospital (Unknown); Euskal Herriko Unibertsitatea. Universidad del Pais Vasco. (Unknown); Osakidetza (Other)
Responsible Party: Juan Bautista Gáldiz, Hospital de Cruces. Osakidetza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV2009111087; GV 2009111087 (Registry Identifier: GV 2009111087)
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: COPD; COPD Exacerbation
Keywords: COPD; Rehabilitation; Neuromuscular stimulation; Quadriceps muscle; Magnetic stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- repetitive neuromuscular stimulation (Experimental): repetitive neuromuscular stimulation of the quadriceps arm are patients actively stimulated at increasing intensity to afford maximal contraction during training sessions
  Interventions: Device: Repetitive magnetic stimulation of the quadriceps muscle

INTERVENTIONS:
Device: Repetitive magnetic stimulation of the quadriceps muscle — During 8 weeks, 7-10 days after hospital release, patients will receive repetitive magnetic stimulation sessions, 15 minutes on each thigh, alternatively two and three days /week.
  Coil location: centered on the union between upper and lower two thirds of the vastus lateralis.
  Stimulation bursts at 10-7 HZ lasting 2 seconds, followed by 4 seconds rest. Intensity will be from 40 to 70% of maximal output, adjusting frequency so that the coil does not overheat, (more than 41ºC).
  Coils are cooled down to 5ºC before sessions.
  Other Names: MEDTRONIC Magpro MCF125; Refrigerated 60mm circular coil.

SUMMARY:
The aims of this study are:1.To evaluate the utility of quadriceps RMNMS (repetitive magnetic neuromuscular stimulation) in the evolution of COPD patients after hospital admission for acute exacerbation.2 To evaluate the time schedule of recovery changes in muscle parameters ,exercise capacity and quality of life after acute exacerbation. 3.To test the use of this new method of training in acute clinical situations. Patients: COPD patients admitted to the Hospital with acute exacerbation. Group 1: RMNMS Treatment .Group 2 : sham RMNMS treatment. Randomized assignment by minimization method. PROTOCOL Training Group: 10 days after discharge and during 8 weeks, 2-3 days/week.

Measures: Spirometry, Plethysmography ,Diffusion Test. Main outcomes: Exercise test (Six minutes walking distance). Muscle function: MVC. Health related quality of life.

DETAILED DESCRIPTION:
Study type Randomized controlled clinical trial with the aim of evaluating an eight-week protocol of repetitive magnetic stimulation (RMNMS) of the quadriceps muscle in COPD patients after inhospital treated exacerbations. The outcomes to be assessed are parameters relating to quadriceps muscle function, exercise capacity (Six minutes walking distance, 6MWD) and quality of life.

Study design and procedures:

Patients will receive information about the investigation, the procedures that will be carried out and their risks, and shall provide written consent in the consent form approved by the Cruces Hospital Ethics and Clinical Trials Committee. Regarding outcome evaluations, all patients, on full intensity and sham RMNMS, will be subjected to identical assessments and functional procedures.

Evaluation for inclusion includes clinical anamnesis and physical exam, chest X-ray evaluation and general blood exam and biochemistry, including creatine kinase (CK) and lactic dehydrogenase (LD). In the week before the start of stimulation treatment and 3 month after hospital discharge, following measurements will be carried out:

* Pulmonary function tests
* Health-related quality of life, using the SF3626 and the Saint George Respiratory Questionnaire(SGRQ), both self administered.
* Body composition: fat-free mass (FFM) using the bioelectric impedance method (Bodystat-500 Bodystat Ltd, Douglas, UK) and expressed as a fat-free mass index (FFMI), which is the result of FFM/(height)2, height expressed in meters.
* Peripheral muscle function: Maximal voluntary contraction of the quadriceps (MVCQ) measured in five maximum isometric contraction efforts (knee-extension attempts) using a Biopac dynamometer (TSD 121C), Biopac system (Biopac System, La Jolla CA, USA) and AcqKnowledge software.
* Six-minute walking test (6MWT): carried out over the same 30 m stretch, according to the standard procedure.(Am J Respir Crit Care Med 2002;166:111e7.) A minimum of three measurements shall be carried out in the initial assessment and two during post-protocol evaluation.

RMNMS training protocol: training sessions will start between 7 and 10 days after hospital discharge.

Patients in the RMNMS group will be subjected to repetitive to magnetic stimulation in sessions of 15 min on each thigh, alternatively two and three days per week, for a period of eight weeks. The assessment is to be repeated three months after hospital discharge.

Stimulation: repetitive magnetic stimulation training of the quadriceps, RMNMS, will be provided by a MEDTRONIC Magpro MCF125 electromagnet with refrigerated circular coils of 60 mm radius, applied at the point between the upper third and the lower two-thirds of the vastus lateralis,the optimum location for eliciting a contraction response,as determined by our volunteer validation study.

Patients will be in sitting or recumbent position with the knee flexed at 90º and the ankle fixed by a strap. The intensity and frequency of stimulation will be adjusted according to the patient's tolerance and the performance of the equipment. Stimulation followed a cyclical pattern of two seconds ON, with contraction elicited by a burst of twitches, and four seconds OFF, repeated over a period of 15 min on each thigh. With the coil being cooled in advance to 5 ºC, it is possible to maintain an initial intensity of 40% of the equipment's maximum stimulation capacity (2 T) at 15 Hz (stimulus per second), ending the protocol at an intensity of 70% at 7 Hz.

Intensity was increased by 5% every two sessions, on the condition that the patient had not reported pain caused by the stimulation or unpleasant sensations following the previous session. In these cases patients will be examined and blood sampled to determine CK and LD determinations.

Control group: patients will received sham training at 20% intensity with same schedule and evaluations as RMNMS patients. Identical to RMNMS patients, the assessment is to be repeated three monts after hospital discharge.

Randomization Patients will be randomized either to intervention group 1, RNMMS or to the sham training control group 2. Scrambling code assignment will be performed and patients will be assigned,using the stratification method considering four factors: age ≥ 65 vs. <65 years, previous admissions yes / no, ≥ 250 vs. walking test < 250 meters and FEV1 ≥ 50 vs. <50%; with this method the aim is to obtain a sufficient representation of these four parameters, both in the control and in the treatment group.

Blinding will be ensured by placing stimulation coils with effective or simulated load in patients and by blinding the outcome assessment that will be conducted without any reference to membership to a specific group. Given the complexity of the design, a triple blind would be unrealistic, so that the therapist himself is familiar with the assignment group. And also to minimize the differences assigned to both groups, we will monitor the treatment and record all incidents that may exist during the process.

Sample size The improvement in distance walked in the 6 minute walking test is regarded as the main variable to evaluate improvement after discharge. An estimated population of 32 patients, sixteen in each arm of the trial would be enough to show an improvement of 50 meters (which is determined as clinically relevant by the various studies and the experience of specialists), with a power of 90% (beta) and a possible significance of 5% (alpha).

Statistical analysis The nonparametric Mann Whitney test will be used for comparison between groups, while Wilcoxon's test for paired data will be used to evaluate the effects of the (training or control) interventions within each group.

Comparison of the inter-group differences will be performed by comparing the percentage change per variable. Correlations between variables will be analysed using Spearman's nonparametric coefficient. Statistical significance: p < 0.05. The 95% confidence interval (CI) will also be provided.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and functional diagnosis of COPD.
* Hospital admission because of COPD exacerbation in respiratory department, ICU or emergency department
* Hospital discharge.

Exclusion Criteria:

* Cardiac pacemaker.
* Exacerbation because of major Heart disease or pulmonary embolism.
* Lung cancer or disseminated neoplasic disease.
* Severe renal or hepatic disease.
* neurological disease, musculoskeletal or cardiovascular or on any treatment that might interfere with the completion of the protocol and the assessment of functional outcomes.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Six minute walking distance | 3 months
  One week after hospital release patients are evaluated and initiate treatment with intense magnetic stimulation or placebo. Measurements are repeated after 3 months.

SECONDARY OUTCOMES:
quality of life CRQ | 3 months
  One week after hospital release patients are evaluated and initiate treatment with intense magnetic stimulation or placebo. Measurements are repeated after 3 months.
Maximal voluntary contraction of the quadriceps | three months
  One week after hospital release patients are evaluated and initiate treatment with intense magnetic stimulation or placebo. Measurements are repeated after 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Cruces, Barakaldo, Bizkaia, Spain

REFERENCES:
- [Background] Coronell C, Orozco-Levi M, Mendez R, Ramirez-Sarmiento A, Galdiz JB, Gea J. Relevance of assessing quadriceps endurance in patients with COPD. Eur Respir J. 2004 Jul;24(1):129-36. doi: 10.1183/09031936.04.00079603. PMID 15293615
- [Background] Barreiro E, Schols AM, Polkey MI, Galdiz JB, Gosker HR, Swallow EB, Coronell C, Gea J; ENIGMA in COPD project. Cytokine profile in quadriceps muscles of patients with severe COPD. Thorax. 2008 Feb;63(2):100-7. doi: 10.1136/thx.2007.078030. Epub 2007 Sep 17. PMID 17875568
- [Background] Bustamante V, Casanova J, Lopez de Santamaria E, Mas S, Sellares J, Gea J, Galdiz JB, Barreiro E. Redox balance following magnetic stimulation training in the quadriceps of patients with severe COPD. Free Radic Res. 2008 Nov;42(11-12):939-48. doi: 10.1080/10715760802555569. PMID 19031320
- [Background] Bustamante V, Lopez de Santa Maria E, Gorostiza A, Jimenez U, Galdiz JB. Muscle training with repetitive magnetic stimulation of the quadriceps in severe COPD patients. Respir Med. 2010 Feb;104(2):237-45. doi: 10.1016/j.rmed.2009.10.001. Epub 2009 Nov 5. PMID 19896353
- [Background] Barreiro E, Peinado VI, Galdiz JB, Ferrer E, Marin-Corral J, Sanchez F, Gea J, Barbera JA; ENIGMA in COPD Project. Cigarette smoke-induced oxidative stress: A role in chronic obstructive pulmonary disease skeletal muscle dysfunction. Am J Respir Crit Care Med. 2010 Aug 15;182(4):477-88. doi: 10.1164/rccm.200908-1220OC. Epub 2010 Apr 22. PMID 20413628